CLINICAL TRIAL: NCT02924649
Title: Early Mobilisation by Head-up Tilt With Stepping Compared With Standard Care After Severe Traumatic Brain Injury - a Randomised Clinical Feasibility Trial
Brief Title: Early Mobilisation After Severe Traumatic Brain Injury
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: University Hospital Bispebjerg and Frederiksberg (Other)
Responsible Party: Principal Investigator, Kirsten Moller, Professor, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-16030775
Record Dates: First submitted 2016-10-03; First posted 2016-10-05 (Estimated); Last update posted 2019-05-24 (Actual); Status verified 2019-05

CONDITIONS: Brain Injuries
Keywords: Brain injury; Early mobilisation; Consciousness; Cerebral blood flow; Blood pressure
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Early Intensive mobilisation (Experimental): As early as possible the experimental group will receive mobilisation on a tilt table for up to 20 minutes 5 days a week for four weeks using an ERIGO tilt table. If orthostatic hypotension occur the patient is moved to supine until parameters are stable again. Hereafter the mobilisation will continue until the patient has completed 20 minutes of standing exercise.
  Interventions: Procedure: Early Intensive mobilisation
- Standard care group (No Intervention): The standard care group will receive daily mobilisation to the seated position.

INTERVENTIONS:
Procedure: Early Intensive mobilisation — The intervention will be performed using a tilt table with integrated stepping movements of the lower extremity (ERIGO, HOCOMA, Switzerland). The goal of the intervention session is that the patient stands upright for 20 minutes. If orthostatic intolerance or increase in intracranial pressure occurs the session will be paused. When the patient is stable mobilization is continued.
  Arms: Early Intensive mobilisation

SUMMARY:
Increasing focus on the negative effects of bed rest have become more apparent in the intensive care unit within the last decade. A few studies have found an association between early rehabilitation starting at the intensive care unit and outcome after discharge from rehabilitation. The early mobilization presents with challenges regarding haemodynamic stability. The aim of this trial is to assess the feasibility before conducting a larger randomised trial that will investigate benefits and harms of an intensive physical rehabilitation intervention focusing on mobilisation to the upright position, starting as early as clinically feasible in the intensive care unit

DETAILED DESCRIPTION:
Patients with severe acquired brain injury (ABI) may benefit from early and intensive rehabilitation that in part consists of physical exercise. Studies have found an association between higher-level physical activities and final outcome in patients with ABI. A higher-level activity for patients with severe ABI and disorders of consciousness consists primarily of mobilization to upright standing position on a tilt-table. Intense higher level activities of severe ABI patients are usually not initiated in the acute stage after injury but rather at a later, sub acute stage (weeks), when the patients have been stabilized and transferred to a highly specialized rehabilitation unit. Andelic et al (2012) conducted a non-randomized cohort study where they investigated the effects of early rehabilitation at the intensive care unit. Although the consistency of the rehabilitation paradigm was unspecified, they did observe a benefit of early intervention. A recent randomized pilot study in 31 patients with acute severe ABI and disorders of consciousness concluded that early mobilization using a tilt-table with integrated stepping that increases the venous return of blood to the heart, could be conducted safely, with significant improvements after three months. The hypothesis that early mobilization of patients with severe traumatic brain injury leads to better functional outcome at discharge from the rehabilitation unit and at one year post injury compared to patients that receive usual care needs to be tested in a larger clinical trial.

In parallel, the physiological changes the patients experience due to their injury and the wast amount of bed rest and the possible association with the patients' clinical outcome are explored. Training is often limited by orthostatic intolerance. The physiological mechanisms causing orthostatic hypotension and their recovery have not been thoroughly investigated. In other patient populations with neurally mediated syncope or orthostatic hypotension, intensive tilt-table training has been shown to be beneficial. In addition, recent studies including a large number of ABI patients have found an association between impaired cerebral autoregulation measured the first days after injury and an unfavorable outcome.

Therefore, we wish to assess the feasibility of an early head-up tilt protocol in patients with severe TBI, not only in terms of the number of patients that are successfully mobilised, but also of the number of adverse events and reactions. In exploratory analyses, we will assess physiological outcomes within the first four weeks and clinical outcomes at three months and one year.

The intervention group receives an early and intensive mobilization programme with head-up tilt, during their stay in the intensive care unit and throughout the early stages of rehabilitation. Mobilization will be conducted using a tilt-table with integrated stepping (The ERIGO® from HOCOMA company in Switzerland). The programme will be conducted as a supplement to the patient's usual care.The tilt-table intervention is applied five times per week for a maximum of four weeks during the stay in the neurointensive care unit. Each session consists of 20 min. mobilization. Within each session the patient will be moved to the tilt-table and secured with straps and harness. The patient is then mobilized step wise to 30°, 50° and 70° head-up tilt in one min. intervals while blood pressure, heart rate, and respiratory rate are closely monitored. Cerebral perfusion pressure and intracranial pressure are monitored if relevant. If at any time the predetermined safety limits for blood pressure, cerebral perfusion pressure, intracranial pressure or heart rate are violated, the patient is lowered to 0° tilt (supine position). This procedure is continued until the patient has been tilted upright for a maximum of 20 min. or until a total duration of 40 min. for the head-up tilt procedure has been reached.

If the patient is discharged from the intensive care unit before four weeks, training will continue at the department of neurorehabilitation with a pre-specified tilt-table protocol consisting of mobilization twice a day on a similar tilt-table. Occasionally patients will be transferred to an intensive care unit at another hospital, while waiting for a further training at the department of neurorehabilitation. These patient will continue their mobilization programme on a regular tilt-table without active stepping. Patients who show functional improvement beyond the scope of tilt-table training (e.g. are able to stand from a chair) before the study period has ended, will have their final evaluation performed immediately hereafter and subsequently the standard rehabilitation regimen will be continued.

The control group receives standard care consisting of interdisciplinary rehabilitation. A very small part of the standard care consists of mobilizing the patient to the edge of the bed or to a wheelchair.

At inclusion the patients will be randomized to either group through an open ended blinded randomization procedure, with stratification according to the patients Glasgow Coma Score at the time (3-6 or 7-10). The randomization will consist of blocks of random sizes.

Assuming that the normality assumption is not violated the functional scores and the physiological data will be analysed with analysis of variance (ANOVA) or other linear regression models that takes into account more than two measures over time. Between-group analysis of demographic data will be performed using Student's t test with unequal variance for analysis of two groups or the chi-square test for nominal data.

ELIGIBILITY:
Inclusion Criteria:

* Traumatic brain injury (TBI)
* Disorders of consciousness (with a tentative diagnosis of the vegetative or minimally conscious state), with a Glasgow Coma Score < 10 during wake-up call.
* Stable intracranial pressure (ICP < 20 mmHg for 24 hours).
* Must be able to mobilise beyond 30 degrees elevation

Exclusion Criteria:

* Unstable fractures contraindicating mobilisation.
* Known heart disease or liver cirrhosis prior to brain injury.
* Spinal cord injury.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility outcome | Within the first four weeks of the study (during the intervention period)
  Successful inclusion of 60% or more of the patients. The intervention will be considered feasible if at least 80% of the intended treatment sessions are applied to at least 70% of the patients.
  Adverse events and reactions (serious and not serious) and suspected unexpected serious adverse reactions

SECONDARY OUTCOMES:
Coma Recovery Scale - Revised (CRS-R) | Measured at inclusion, after four weeks, three months and at one year follow-up
Early Functional Ability (EFA) | Measured at inclusion, after four weeks, three months and at one year follow-up
  The Early Functional ability scale measures the gap between FIM and the Glasgow Coma Score.
Functional Independence Measures (FIM) | Measured at inclusion, after four weeks, three months and at one year follow-up
Autoregulation of cerebral blood flow | At baseline, after two weeks and at four weeks
  Using Transcranial Doppler and mean arterial pressure two express cerebral autoregulation during mobilisation to standing position. At these points we will measure carbon dioxide partial pressure and heart rate.
Time with post-traumatic amnesia (PTA) | Duration of posttraumatic amnesia
  The neuro psychologists at the departments are assessing this point on a regular basis
Length of stay at the Neurointensive Care Unit and the Rehabilitation department | Duration of length of stay
  Length of stay measured in days

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten Møller, Professor, Study Director — Rigshospitalet, Dept. of anaesthesiology, Rigshospitalet
Locations (1):
- Rigshospitalet,, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Horn SD, DeJong G, Smout RJ, Gassaway J, James R, Conroy B. Stroke rehabilitation patients, practice, and outcomes: is earlier and more aggressive therapy better? Arch Phys Med Rehabil. 2005 Dec;86(12 Suppl 2):S101-S114. doi: 10.1016/j.apmr.2005.09.016. PMID 16373145
- [Background] DeJong G, Hsieh CH, Putman K, Smout RJ, Horn SD, Tian W. Physical therapy activities in stroke, knee arthroplasty, and traumatic brain injury rehabilitation: their variation, similarities, and association with functional outcomes. Phys Ther. 2011 Dec;91(12):1826-37. doi: 10.2522/ptj.20100424. Epub 2011 Oct 14. PMID 22003165
- [Background] Riberholt CG, Thorlund JB, Mehlsen J, Nordenbo AM. Patients with severe acquired brain injury show increased arousal in tilt-table training. Dan Med J. 2013 Dec;60(12):A4739. PMID 24355448
- [Background] Wilson BA DS, Tunnard C, Watson P and Florschutz G. The Effect of Positioning on the Level of Arousal and Awareness in Patients in the Vegetative State or the Minimally Conscious State: A Replication and Extension of a Previous Finding. BRAIN IMPAIRMENT. 2013;14(3):475-9.
- [Background] Elliott L, Coleman M, Shiel A, Wilson BA, Badwan D, Menon D, Pickard J. Effect of posture on levels of arousal and awareness in vegetative and minimally conscious state patients: a preliminary investigation. J Neurol Neurosurg Psychiatry. 2005 Feb;76(2):298-9. doi: 10.1136/jnnp.2004.047357. No abstract available. PMID 15654064
- [Background] Newman M, Barker K. The effect of supported standing in adults with upper motor neurone disorders: a systematic review. Clin Rehabil. 2012 Dec;26(12):1059-77. doi: 10.1177/0269215512443373. Epub 2012 May 29. PMID 22643724
- [Background] Andelic N, Bautz-Holter E, Ronning P, Olafsen K, Sigurdardottir S, Schanke AK, Sveen U, Tornas S, Sandhaug M, Roe C. Does an early onset and continuous chain of rehabilitation improve the long-term functional outcome of patients with severe traumatic brain injury? J Neurotrauma. 2012 Jan 1;29(1):66-74. doi: 10.1089/neu.2011.1811. Epub 2011 Dec 5. PMID 21864138
- [Background] Frazzitta G, Valsecchi R, Zivi I, Sebastianelli L, Bonini S, Zarucchi A, Matteri D, Molatore K, Maestri R, Saltuari L. Safety and Feasibility of a Very Early Verticalization in Patients With Severe Traumatic Brain Injury. J Head Trauma Rehabil. 2015 Jul-Aug;30(4):290-2. doi: 10.1097/HTR.0000000000000135. No abstract available. PMID 26147317
- [Background] Riberholt CG, Olesen ND, Thing M, Juhl CB, Mehlsen J, Petersen TH. Impaired Cerebral Autoregulation during Head Up Tilt in Patients with Severe Brain Injury. PLoS One. 2016 May 11;11(5):e0154831. doi: 10.1371/journal.pone.0154831. eCollection 2016. PMID 27168188
- [Background] Verheyden B, Ector H, Aubert AE, Reybrouck T. Tilt training increases the vasoconstrictor reserve in patients with neurally mediated syncope evoked by head-up tilt testing. Eur Heart J. 2008 Jun;29(12):1523-30. doi: 10.1093/eurheartj/ehn134. Epub 2008 Mar 27. PMID 18375398
- [Background] Lang EW, Lagopoulos J, Griffith J, Yip K, Mudaliar Y, Mehdorn HM, Dorsch NW. Noninvasive cerebrovascular autoregulation assessment in traumatic brain injury: validation and utility. J Neurotrauma. 2003 Jan;20(1):69-75. doi: 10.1089/08977150360517191. PMID 12614589
- [Background] Liu X, Czosnyka M, Donnelly J, Budohoski KP, Varsos GV, Nasr N, Brady KM, Reinhard M, Hutchinson PJ, Smielewski P. Comparison of frequency and time domain methods of assessment of cerebral autoregulation in traumatic brain injury. J Cereb Blood Flow Metab. 2015 Feb;35(2):248-56. doi: 10.1038/jcbfm.2014.192. Epub 2014 Nov 19. PMID 25407266
- [Background] Giacino JT, Kalmar K, Whyte J. The JFK Coma Recovery Scale-Revised: measurement characteristics and diagnostic utility. Arch Phys Med Rehabil. 2004 Dec;85(12):2020-9. doi: 10.1016/j.apmr.2004.02.033. PMID 15605342
- [Background] Hankemeier A, Rollnik JD. The Early Functional Abilities (EFA) scale to assess neurological and neurosurgical early rehabilitation patients. BMC Neurol. 2015 Oct 19;15:207. doi: 10.1186/s12883-015-0469-z. PMID 26482349
- [Background] van Baalen B, Odding E, van Woensel MP, Roebroeck ME. Reliability and sensitivity to change of measurement instruments used in a traumatic brain injury population. Clin Rehabil. 2006 Aug;20(8):686-700. doi: 10.1191/0269215506cre982oa. PMID 16944826
- [Background] Stubbs PW, Pallesen H, Pedersen AR, Nielsen JF. Using EFA and FIM rating scales could provide a more complete assessment of patients with acquired brain injury. Disabil Rehabil. 2014;36(26):2278-81. doi: 10.3109/09638288.2014.904935. Epub 2014 Mar 28. PMID 24678931
- [Background] Gronwall D, Wrightson P. Duration of post-traumatic amnesia after mild head injury. Journal of Clinical Neuropsychology. 1980;2(1):51-60.
- [Background] Imholz BP, Wieling W, van Montfrans GA, Wesseling KH. Fifteen years experience with finger arterial pressure monitoring: assessment of the technology. Cardiovasc Res. 1998 Jun;38(3):605-16. doi: 10.1016/s0008-6363(98)00067-4. PMID 9747429
- [Background] Giller CA, Bowman G, Dyer H, Mootz L, Krippner W. Cerebral arterial diameters during changes in blood pressure and carbon dioxide during craniotomy. Neurosurgery. 1993 May;32(5):737-41; discussion 741-2. PMID 8492848
- [Background] Beninato M, Gill-Body KM, Salles S, Stark PC, Black-Schaffer RM, Stein J. Determination of the minimal clinically important difference in the FIM instrument in patients with stroke. Arch Phys Med Rehabil. 2006 Jan;87(1):32-9. doi: 10.1016/j.apmr.2005.08.130. PMID 16401435
- [Derived] Riberholt CG, Olsen MH, Berg RMG, Mehlsen J, Moller K. Dynamic cerebral autoregulation during early orthostatic exercise in patients with severe traumatic brain injury: Further exploratory analyses from a randomized clinical feasibility trial. J Clin Neurosci. 2021 Oct;92:39-44. doi: 10.1016/j.jocn.2021.07.047. Epub 2021 Aug 3. PMID 34509259
- [Derived] Riberholt CG, Olsen MH, Sondergaard CB, Gluud C, Ovesen C, Jakobsen JC, Mehlsen J, Moller K. Early Orthostatic Exercise by Head-Up Tilt With Stepping vs. Standard Care After Severe Traumatic Brain Injury Is Feasible. Front Neurol. 2021 Apr 14;12:626014. doi: 10.3389/fneur.2021.626014. eCollection 2021. PMID 33935935
- [Derived] Riberholt CG, Lindschou J, Gluud C, Mehlsen J, Moller K. Early mobilisation by head-up tilt with stepping versus standard care after severe traumatic brain injury - Protocol for a randomised clinical feasibility trial. Trials. 2018 Nov 8;19(1):612. doi: 10.1186/s13063-018-3004-x. PMID 30409170